CLINICAL TRIAL: NCT03637127
Title: Acute Exposure to Hypoxia in Precapillary Pulmonary Hypertension: Physiological and Clinical Effects at Rest and During Exercise
Brief Title: Acute Exposure of Simulated Hypoxia on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00455_A4
Record Dates: First submitted 2018-07-09; First posted 2018-08-17 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Hypertension
Keywords: Simulated altitude; cognitive function
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Including a baseline assessment and assessments under simulated altitude and normoxia.
Who Masked: Participant
Masking Description: The allocated gas mixture will not be disclosed to the patient since he will breath through a facemask during both interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order air-hypoxia (Experimental): The participants will be exposed to shamed hypoxia (FiO2: 20.9% equivalent to sea level and consecutively to simulated altitude (FiO2: 15.1% equivalent to 2500m above sea level) administered by an altitude Simulator ("Altitrainer, SMTEC"), simulated altitude (FiO2: 15.1%), with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1%); Device: Shamed Hypoxia (FiO2: 20.9)
- Order hypoxia-air (Experimental): The participant will be exposed to hypoxia (FiO2, 15.1% equivalent to 2500m above sea level), simulated altitude (FiO2: 15.1%), and consecutively to shamed hypoxia (FiO2, 20.9%) administered by an altitude simulator ("Altitrainer, SMTEC") with a facemask.
  Interventions: Device: Simulated Altitude (FiO2: 15.1%); Device: Shamed Hypoxia (FiO2: 20.9)

INTERVENTIONS:
Device: Simulated Altitude (FiO2: 15.1%) — Inhalation of deoxygenated air through a altitude simulator ("Altitrainer"), for approx. 1 hour. given by a facemask.
Device: Shamed Hypoxia (FiO2: 20.9) — Inhalation of unmodified air through an altitude Simulator ("Altitrainer") for approximately 1 hour given by a facemask

SUMMARY:
Randomized crossover Trial in patients with Pulmonary Hypertension (PAH, CTEPH) to assess the acute response to simulated altitude (FiO2:15.1, equivalent to 2500m above sea level) on cognitive functions.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Zurich (460m asl) including Echocardiography, Right heart catheterization, six-minute walk test (6MWT), pulmonary function test, clinical assessment and blood gas Analysis.

Randomly assigned to the order of testing, the participants will be tested under simulated altitude (FiO2: 15.1% with the "AMC Altitrainer") and shamed altitude with the same device.

During the exposure to simulated altitude (FiO2: 15.1%) of approximately 1 hour, the participants will perform cognitive function test .

The results will be compared under hypoxic and normal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* PH diagnosed according to internation Guidelines: mean pulmonary artery pressure (mPAP) ≥ 25 mmHg along with a pulmonary artery wedge pressure (PAWP) ≤15 mmHg during right heart catheterization at the time of initial diagnosis
* PH class 1 (PAH) or 4 (CTEPH)
* Stable condition, on the same medication for > 4 weeks
* Patient live permanently at an altitude < 1000m asl.

Exclusion Criteria:

* Resting partial oxygen pressure (PaO2) ≤7.3 kilopascal (kPA) corresponding to the requirement of long-term oxygen therapy > 16hour daily (nocturnal oxygen therapy alone is allowed)
* Severe daytime hypercapnia (pCO2 > 6.5 kPa)
* Susceptibility to high altitude related diseases (AMS, high-altitude pulmonary edema (HAPE), etc.) based on previous experienced discomfort at altitudes.
* Exposure to an altitude >1500m for ≥3 nights during the last 4 weeks before the study participation
* Residence > 1000m above sea level
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with walking disability
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Function test | 2 hours
  Change in cognitive function test time during the exposure to simulated altitude (FiO2: 15.1%) and normoxia

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof., Principal Investigator — University of Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland